CLINICAL TRIAL: NCT00087919
Title: Defining an Obesity QTL on Chromosome 3q
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1263; R01HL074166 (NIH)
Record Dates: First submitted 2004-07-15; First posted 2004-07-19 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maywood: The were 743 subjects were sampled from Maywood, Il. There was no intervention.
- Nigeria: There were 1188 Nigerian sampled from Igbo-Ora and Ibadan, Nigeria. There was no intervention.

SUMMARY:
To investigate the genetic basis of obesity by fine mapping an obesity quantitative trail linkage (QTL) linked to chromosome 3q.

DETAILED DESCRIPTION:
BACKGROUND:

In the last several decades obesity has emerged as a major public health threat. While prevention through lifestyle change is the only long-term solution, better understanding of the physiologic mechanisms would greatly assist development of drugs and targeted prevention. Obesity is a highly heritable condition and while genes must account for a substantial proportion of individual susceptibility they have eluded detection. Powerful new genetic and genomic tools now permit comprehensive evaluation of candidate genes, including all genes under linkage peaks. These tools include new genomic resources (the human genome sequence, databases of common SNPs, and the haplotype map), rapid and inexpensive discovery and genotyping and new analytic methods (haplotype-based association and admixture mapping).

DESIGN NARRATIVE:

In a large African American family set Dr. Zhu and colleagues have obtained strong linkage evidence for obesity on chromosome 3q (combined LOD score = 3.7). A prime candidate (adiponectin) lies near this peak. They propose to follow up that finding by combining the epidemiologic data with high-throughput genotyping and move from linkage to association analysis. The results for this QTL will be evaluated within the available environmental factors to assess potential gene-environment and gene-gene interactions. The available phenotypes include body composition, resting metabolic rate, physical activity, plasma insulin, glucose, and leptin. In a family-based design they will examine the linkage peak centered on position 188 cM on chromosome 3q (20 Cm 1-LOD support interval), with the following step-wise strategy: (a) Genotype 200 single nucleotide polymorphisms (SNPs) in this region on 300 families (1,000 individuals); (b) Conduct linkage, linkage disequilibrium and admixture mapping to potentially further narrow the region; and (c) Conduct resequencing and haplotype-based association studies for all candidate genes under the peak. Statistical analysis incorporating intermediate phenotypes and environmental covariates will be used to characterize potential gene x gene or gene x environment interactions. Replication will be tested in additional populations of African and European origin.

ELIGIBILITY:
The survey enrolled a representative random sample of the population the age of 18 and 74, regardless of obesity phenotype.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maywood cohort DNA samples were obtained from a larger cohort of families enrolled in the studies of blood pressure at Loyola University in Maywood, IL. The survey enrolled a representative random sample of the population between the ages of 18 and 74, regardless of obesity phenotype. A subcohort of 775 unrelated participants was selected and oversampled at the upper and lower ends of the BMI distribution to increase the power.
  Nigerian cohort Study participants were recruited from Igbo-Ora and Ibadan in southwest Nigeria as part of a long-term study on the environmental and genetic factors underlying hypertension. The sample comprised 1098 unrelated adults with normal or elevated blood pressure and 155 unrelated participants from Ibadan with elevated blood pressure recruited as controls in the Africa-America Diabetes Mellitus (AADM) study.
Sampling Method: Probability Sample
Enrollment: 1931 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhu, Principal Investigator — Case Western Reserve University